CLINICAL TRIAL: NCT07012889
Title: Safety and Efficacy of Intraoperative Continuous Lidocaine Infusion in Patients Undergoing Laparoscopic Liver Surgery: Effects on Postoperative Pain, Gut Function and Insulin Resistance
Brief Title: Intraoperative Continuous Lidocaine Infusion in Laparoscopic Liver Surgery
Acronym: ICLIL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KB/23/2025
Record Dates: First submitted 2025-04-23; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain After Laparoscopic Liver Resection
Keywords: postoperative pain; laparoscopic liver surgery; lidocaine infusion
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The lidocaine group (Experimental)
  Interventions: Drug: lidocaine infusion
- The placebo group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: lidocaine infusion — The lidocaine group will receive initial intravenous bolus dose of 1.5mg/kg lidocaine over 10 min, followed by a continuous infusion of 1.5 mg/kg/h lidocaine until the end of surgery. The dose of lidocaine will be calculated according to ideal body weight. The placebo group will be administered normal saline at the same volume, infusion rate and timing.
  Arms: The lidocaine group
Other: Placebo — The placebo group will be administered normal saline 0.9% at the same volume, infusion rate and timing as lidocaine in the lidocaine group
  Arms: The placebo group

SUMMARY:
The goal of this clinical trial is to learn about effect of intraoperative continuous lidocaine infusion on postoperative pain, gut function and insulin resistance in patients undergoing laparoscopic liver surgery in adults. It will also learn about the safety of this infusion in this setting. The main questions it aims to answer are: does the intraoperative continuous systemic lidocaine infusion lower the opioid consumption 24h after surgery? Is the time to first flatus after surgery reduced? Is there increases in insulin resistance after intraoperative lidocaine infusion? Researchers will compare intraoperative continuous systemic lidocaine infusion to a placebo (a look-alike substance that contains no drug, which will be normal saline administered at the same volume, infusion rate and timing) to see if intraoperative continuous systemic lidocaine infusion reduces postoperative pain after laparoscopic liver resection.

Participants will receive intraoperative continuous systemic lidocaine infusion or placebo. Clinical assessment will be based on gathering data of NRS scores after the surgery, time to first flatus or stool. How much opioids the patients need in the first 3 postoperative days. Laboratory assessment will include the evaluation of fasting blood glucose concentration and insulin levels preoperatively and on 1, 2 and 3 postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old
* patients scheduled for laparoscopic liver surgery
* patients classified as American Society of Anesthesiology (ASA) physical status I- III

Exclusion Criteria:

* medical history of seizure disorders
* allergy to Lidocaine
* cardiac rhythm disorders (e.g. sick sinus syndrome, Adams-Stockes syndrome, II- and III-degree AV blocks, double- bundle branch block, HR < 50/min)
* systolic heart failure (ejection fraction <50%)
* hepatic dysfunction (aspartate aminotransferase or alanine transaminase or total bilirubin >2.5 times the upper limit of normal)
* renal impairment (GFR < 50ml/min/1.73 m2)
* weight less than 45 kg, BMI > 30
* metastases occurring in other distant organs
* recent use of any analgesic medication within 48h before surgery
* history of alcohol or substance abuse
* chronic pain syndrome
* chronic opioid use
* inability to comprehend NRS or complete questionnaires due to language barrier or cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-03-02 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
opioid consumption during the first 24 hours after the surgery | First 24 hours after the end of the surgery (extubation)
  the mean cumulative opioid consumption during the first 24 hours after the surgery

SECONDARY OUTCOMES:
gut recovery | from the end of the surgery (extubation) until the date of first documented flatus or stool, whichever came first, assessed up to 72 hours
  time to first flatus or stool after surgery
HOMA-IR | from the day 0 after surgery to day 3 after surgery
  fasting blood glucose concentration, insulin levels preoperatively